CLINICAL TRIAL: NCT06302075
Title: Evaluation of Functional Recovery of Patients Undergoing Medial Monocompartmental Knee Prosthesis With One Day Protocol Versus Fast Protocol
Brief Title: Functional Recovery After Medial Monocompartmental Knee Prosthesis: One Day Protocol Versus Fast Protocol
Acronym: UKA-L2086
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKA-L2086
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Gonarthrosis
Keywords: Gonarthrosis; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One Day Rehabilitation (Experimental): discharged home the day after the operation (24 hours) and carrying out outpatient rehabilitation according to the clinical standard
  Interventions: Other: One Day Rehabilitation
- Fast Rehabilitation (Active Comparator): discharged to the rehabilitation department of the Institute 48 hours after surgery which carries out rehabilitation during the hospital stay according to the clinical standard
  Interventions: Other: Fast Rehabilitation

INTERVENTIONS:
Other: One Day Rehabilitation — Patient discharged at home the day after the operation and carrying out outpatient rehabilitation according to the clinical standard
  Arms: One Day Rehabilitation
Other: Fast Rehabilitation — Patient discharged to the rehabilitation department of the Institute 48 hours after surgery which carries out rehabilitation during the hospital stay according to the clinical standard
  Arms: Fast Rehabilitation

SUMMARY:
The study is defined as prospective, randomized, interventional single-center; the general aim is to evaluate the post-operative recovery of the patient who carries out rehabilitation with the one day protocol (Group A), compared to the patient who carries out rehabilitation during the hospital stay with the fast protocol (group B).

DETAILED DESCRIPTION:
The study is defined as prospective, randomized, interventional single-center; the general aim is to evaluate the post-operative recovery of the patient who carries out rehabilitation with the one day protocol (Group A), compared to the patient who carries out rehabilitation during the hospital stay with the fast protocol (group B).

The difference will be evaluated with the Knee Society Scopre (KSS) questionnaire at 1 month after the operation.

The population is made up of two groups of patients:

25 patients Group A: one day protocol; experimental group discharged home the day (24h) after the operation and carrying out rehabilitation according to the clinical standard 25 patients Group B: fast protocol; control group discharged to the rehabilitation department of the Institute 48 hours after surgery which carries out rehabilitation during the hospital stay according to the clinical standard

The subjects will undergo the following assessments:

* Pre-admission
* Knee replacement surgery
* Rehabilitation
* Questionnaires and evaluation scales at 7 and 15 days (+/- 2 days), at 1, 3, 6 months (+/- 7 days) and 12 months (+/- 1 month) after surgery. If necessary, they can be collected by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age 40<x<85 included
* Medial monocompartmental gonarthrosis grade 3-4 sec Kellgren-Lawrence
* Primary medial gonarthrosis
* Signing of the Informed Consent and consent to collaborate in all study procedures.

Exclusion Criteria:

* Cognitive decline
* Psychiatric disorders
* Neuromuscular disorders
* Age > 85 years or <40
* Lateral gonarthrosis grade 3-4 sec Kellgren-Lawrence
* Patella symptoms
* Secondary medial gonarthrosis
* Minor age
* Pregnant women (self-declaration)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) from 0 to 100 (whether higher scores mean a better outcome) | 1 month
  To evaluate the KSS at 1 month from the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico San Siro, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided